CLINICAL TRIAL: NCT01736579
Title: A Study of the Long-Term Safety and Efficacy of Immune Globulin Intravenous (Human), 10% Solution (IGIV, 10%) in Mild to Moderate Alzheimer´s Disease
Brief Title: Long-Term Study of IGIV, 10% in Alzheimer´s Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated because the first Phase 3 did not demonstrate efficacy on the co-primary endpoints. The known safety profile remained unchanged.
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 161202
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer´s Disease
MeSH Terms: interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IGIV, 10% at 0.2 g/kg body weight (Experimental): IGIV, 10% at 0.2 g/kg body weight every 2 weeks for up to 3 years, 6 months.
  Interventions: Drug: Immune Globulin Intravenous (Human), 10% (IGIV, 10%)
- IGIV, 10% at 0.4 g/kg body weight (Experimental): IGIV, 10% at 0.4 g/kg body weight every 2 weeks for up to 3 years, 6 months
  Interventions: Drug: Immune Globulin Intravenous (Human), 10% (IGIV, 10%)

INTERVENTIONS:
Drug: Immune Globulin Intravenous (Human), 10% (IGIV, 10%)
  Other Names: Gammagard Liquid

SUMMARY:
The purpose of this long-term study is to provide additional evidence of safety and efficacy of IGIV, 10% treatment in participants with Alzheimer´s Disease who have completed the Phase 3 Baxter precursor study 160701. All participants will receive IGIV, 10% at either 0.2 g/kg or 0.4 g/kg body weight depending on their treatment assignment in Baxter study 160701. Participants and investigators will be blinded to dose unless otherwise notified by the sponsor.

ELIGIBILITY:
Main Inclusion Criteria:

* Completed 18 months of study treatment and assessments in Baxter precursor study 160701
* Diagnosis of probable Alzheimer´s Disease (AD)
* Able to comply with testing and infusion regimen (including adequate corrected visual acuity and hearing ability)
* Has a caregiver (study partner) who is willing and able to participate

Main Exclusion Criteria:

* Significant neurological disease other than AD
* Clinically significant cardiac/cardiovascular problems (e.g. uncontrolled blood pressure, atrial fibrillation, heart disease, clotting disorders, strokes, or recent heart attack)
* Contraindication to undergoing MRI (e.g. pacemaker [with the exception of an MRI-compatible pacemaker], severe claustrophobia, ferromagnetic implants such as a metal plate)
* Specific findings on brain MRI (microhemorrhages, superficial siderosis, vasogenic edema, a macrohemorrhage, major stroke, or multiple lacunae)
* Active malignancy or history of malignancy within 5 years prior to screening with the exception of the following: adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and stable prostate cancer not requiring treatment
* Uncontrolled major depression, psychosis, or other major psychiatric disorder(s)
* Poorly controlled diabetes
* Serious problems with liver or kidneys
* Known history of hypersensitivity following infusions of human blood or blood components (e.g. human immunoglobulins or human albumin)
* Current or recent treatment with immunomodulatory therapies (with the exception of immunoglobulin and non-systemic and low-dose systemic corticosteroids)
* Recent use of investigational drugs or biologics, including those aimed at altering AD progression (with the exception of immunoglobulin)
* Active immunization for the treatment of AD at any time

There are reasons why it might not be appropriate to participate in this trial. Please contact Medical Information at medinfo@baxter.com for details.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11-29 (Actual); Primary Completion 2013-06-04 (Actual); Study Completion 2013-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at one clinical site in the US.
Pre-assignment Details: Six participants were enrolled (i.e. signed informed consent form), of which 2 failed screening and 4 were treated with study product.
Groups:
- IGIV, 10% at 0.2 g/kg Body Weight: IGIV, 10% at 0.2 g/kg body weight every 2 weeks
- IGIV, 10% at 0.4 g/kg Body Weight: IGIV, 10% at 0.4 g/kg body weight every 2 weeks
Period: Overall Study
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Termination of Study by Sponsor | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: 6 months
Measure: Number; unit: adverse events
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 2 | 2
adverse events
  Non-serious AEs-Mild | 2 | 0
  Non-serious AEs-Moderate | 1 | 1
  SAEs | 0 | 0

2. Primary Outcome: Number of Infusions Temporally Associated With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: 6 months
Measure: Number; unit: infusions
Units Other Than Participants: Infusions
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 2 | 2
Number analyzed (Infusions) | 10 | 7
infusions | 1 | 0

3. Primary Outcome: Number of Infusions Causally Associated With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: 6 months
Measure: Number; unit: infusions
Units Other Than Participants: Infusions
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 2 | 2
Number analyzed (Infusions) | 10 | 7
infusions | 1 | 1

4. Primary Outcome: Number of Infusions Discontinued, Slowed or Interrupted Due to an Adverse Event (AE) or Serious Adverse Event (SAE)
Time Frame: 6 months
Measure: Number; unit: infusions
Units Other Than Participants: Infusions
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 2 | 2
Number analyzed (Infusions) | 10 | 7
infusions | 0 | 0

5. Secondary Outcome: Total Score of the Cognitive Subscale of the Alzheimer's Disease Assessment Scale (ADAS-Cog)
Description: The ADAS-Cog is a validated psychometric instrument that evaluates memory (word recall, word recognition), attention, reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing letter in envelope) and constructional praxis (copying geometric designs). This test was administered by experienced raters certified by Alzheimer's Disease Cooperative Study (ADCS) at the site. Scores on the ADAS-Cog range from 0-70 with higher scores indicating greater impairment.
Time Frame: 6 months
Population: This study was terminated early. Summary tables were not provided for this outcome measure due to the small number of participants (up to 2 participants per arm) because of concerns about patient confidentiality.
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Total Score of the Cognitive Subscale of the Severe Impairment Battery (SIB)
Description: The SIB is a 40-item psychometric assessment that is composed of simple one-step commands combined with gestures. The scoring range is from 0 to 100 with a lower score indicating greater cognitive impairment.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Alzheimer's Disease Cooperative Study (ADCS) - Activities of Daily Living (ADL) Inventory (ADCS-ADL/ ADCS-ADL-severe)
Description: The ADCS-ADL scale is a validated tool to assess instrumental and basic activities of daily living based on a 23 item structured interview of the caregiver or qualified study partner. Scores on the ADCS-ADL range from 0-78 with lower scores indicating greater impairment; hence decreases from baseline reflect potential functional deterioration.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mini Mental State Examination (MMSE)
Description: The MMSE is a test for cognitive dysfunction. The test provides a 30-point composite rating for spatial and temporal orientation, verbal recall, simple attention, working memory, naming, repetition, comprehension, writing and constructional abilities. The total score can range from 0 to 30 with a higher score indicating better function.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Neuropsychiatric Inventory (NPI) Score
Description: The NPI is a validated instrument used to assess behavioral psychopathology in Alzheimer's Disease; it evaluates the frequency and severity of 12 neuropsychiatric features including delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability/lability, apathy, aberrant motor activity, sleep and night-time behavior change, and appetite and eating change. The NPI total score ranged 0-144, with higher scores indicating greater impairment.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Logsdon Quality of Life in Alzheimer's Disease (QOL-AD)
Description: The QOL-AD is a validated, 13-item instrument developed specifically for individuals with dementia. The assessment rates the participant's quality of life for physical, emotional, interpersonal, and environmental domains. The QOL-AD total score ranged 13-52. Lower scores on the QOL-AD are associated with a lower quality of life.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: EQ-5D Questionnaire (Proxy Version)
Description: EQ-5D is a participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome. The EQ-5D also includes a standard vertical 20 cm visual analogue scale (VAS) ranging from best imaginable health state [100] to worst imaginable health state [0]. Caregivers are asked to describe how they believe a participant would rate his/her health state that day.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Healthcare Resource Utilization Questionnaire (HRUQ)
Description: The HRUQ determines if there is a difference in healthcare utilization and health-related expenditures, most notably nursing home (ie, skilled nursing facility) admissions, when subjects are treated with study product. This assessment is performed with the primary caregiver. This assessment is descriptive and does not contain specific scores.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Caregiver Burden Questionnaire
Description: The Caregiver burden questionnaires is a self-administered questionnaire that has been developed to measure the emotional, physical, and social impact of caregiving on Alzheimer's Disease caregivers. A Total score is calculated from this measure by summing the responses across the items. The Total score may range from 9-45, with higher scores indicating greater burden.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Time to Skilled Nursing Facility Placement
Description: Time to skilled nursing facility placement is defined as permanent admission to a skilled nursing facility. Time will be defined as the number of months between enrollment into this clinical study and placement in a skilled nursing facility placement.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Volumetric MRI
Description: Volumetric MRI measurements were obtained to assess rate of whole brain atrophy and ventricular enlargement. Additional volumetric measurements may be analyzed when specific hypotheses and methods are defined. Additional volumetric MRI analysis may include (but may not be limited to) one or more of the following: rate of hippocampal atrophy, entorhinal cortical thickness, and/or regional cortical thinning.
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period (6 months)
Arm/Group | IGIV, 10% at 0.2 g/kg Body Weight | IGIV, 10% at 0.4 g/kg Body Weight
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGIV, 10% at 0.2 g/kg Body Weight (N=2) | IGIV, 10% at 0.4 g/kg Body Weight (N=2)
Infusion Site Pain (General disorders) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Blood Pressure Increased (Investigations) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was an extension of study 160701 and was stopped early due to lack of evidence of clinical benefit of IGIV treatment in Alzheimer's Disease patients in Baxalta study 160701. Summary tables available for safety data only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 12 months after study completion. Baxalta requires a review of results communications (eg, for confidential information) ≥30 days prior to submission or communication. Baxalta may request an additional delay of ≤60 days eg, for intellectual property protection.